CLINICAL TRIAL: NCT00242502
Title: A Phase II Study of the Combination of Bevacizumab and Erlotinib in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Efficacy and Safety Study of Bevacizumab and Erlotinib to Treat Primary Liver Cancer That Cannot be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0874
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-03

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Hepatocellular Carcinoma; Liver Cancer; Bevacizumab; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Erlotinib Hydrochloride; OSI-774; Tarceva; Erlotinib; Avastin
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Erlotinib (Experimental): Bevacizumab 10 mg/kg intravenous every 14 days, repeat cycle every 28 days; Erlotinib 150 mg orally every day continuous dosing.
  Interventions: Drug: Bevacizumab (Avastin); Drug: Erlotinib

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — 10 mg/kg IV every 14 days, repeat cycle every 28 days
  Other Names: Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Erlotinib — 150 mg orally every day continuous dosing, repeat cycle every 28 days
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva

SUMMARY:
The primary objective will be to assess progression-free survival (PFS) measured at 16 weeks following initiation of therapy with the combination of Avastin and erlotinib in patients with unresectable hepatocellular carcinoma (HCC). Progression-free survival is defined as the time from initiation of therapy until documented disease progression or death.

Secondary objectives include: response rate, median and overall survival, toxicity and tolerability, and to ascertain whether there is any correlation of response with prior treatment status and underlying HCC risk factor(s).

DETAILED DESCRIPTION:
Liver cancer growth may be affected by a protein in the body called "vascular epidermal growth factor" (VEGF). A drug that blocks VEGF may be an effective treatment for liver cancer. Avastin is designed to block VEGF. Erlotinib hydrochloride is an investigational drug believed to work on cancer cells by affecting epidermal growth factor receptor (EGFR), a protein that is important to cancer growth.

If the screening evaluations show you are eligible to take part in the study, you may begin treatment. You will receive treatment in 28-day periods called "cycles". Treatment will be given on an outpatient basis. Because this is a research study, the Avastin infusion must be given every time at M. D. Anderson. Because erlotinib hydrochloride is given by mouth, you may take it away from M. D. Anderson.

You will receive Avastin through a needle in a vein on Days 1 and 15 of each cycle. The first dose of Avastin will be given over about 90 minutes. If you do not have a reaction (such as fever/chills), the next dose will be given over about 60 minutes. If again no reaction occurs, each dose after that will be given over about 30 minutes. If you experience a reaction to the Avastin infusion, you may be given acetaminophen (such as Tylenol) by mouth and/or an antihistamine by vein over 30 minutes before each dose to help decrease the risk of further reactions.

You will take erlotinib hydrochloride tablets by mouth every day. It is recommended that erlotinib hydrochloride be taken in the morning with a glass of water. Erlotinib hydrochloride should be taken at least 1 hour before or 2 hours after you have any food, grapefruit juice, vitamins, iron supplements, or other non-prescription medicines.

Before each new cycle of study treatment, you will have urine collected, and blood will be drawn (about 3 tablespoons) for routine blood tests and to check your blood clotting. You will be asked questions about any side effects you may have had and about any medications you are currently taking or have taken since you last saw the study doctor. You will have a complete physical exam, including measurements of vital signs and weight. You will be asked about your ability to perform everyday tasks.

You will also have CT and/or MRI scans of the tumor(s) every 8 weeks. Additional tests may be done during the study if your doctor feels it is necessary for your care. All testing and evaluations must be done at M. D. Anderson.

If you experience severe side effects, treatment may be delayed, stopped, or you may receive smaller doses of the treatment. You may continue to receive study treatment unless the disease gets worse, the side effects are too severe, you decide not to take part any longer, or your doctor decides it is in your best interest to stop treatment. There is no maximum number of cycles that you can receive.

When you stop study treatment, you will be asked to have tests and evaluations done at an end-of-study visit. You will have urine collected, and blood will be drawn (about 3 tablespoons) for routine blood tests and to check your blood clotting. You will be asked questions about any side effects you may have had and about any medications you are currently taking or have taken since you last saw the study doctor. You will have a complete physical exam, including measurements of blood pressure, pulse, temperature, and weight. You will be asked about your ability to perform everyday tasks. You will also have CT and/or MRI scans of the abdomen and pelvis to check on your cancer.

Once you stop receiving study treatment, the study doctor or nurse will continue to check how you are doing, either in the clinic or by telephone if you stop coming to M. D. Anderson, every 3 months for the rest of your life.

This is an investigational study. Erlotinib hydrochloride is approved by the FDA for treatment of lung cancer, but it is not approved for liver cancer, so its use is considered experimental in this study. Avastin is approved by the FDA for treatment of colon and rectal cancer, but it is not approved for the treatment of liver cancer, so its use is considered experimental in this study. Up to 60 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed hepatocellular carcinoma not amenable to curative resection.
2. Patients must have measurable disease as per the Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
3. Patients are allowed to have had up to one prior systemic therapy, including chemotherapy or hormonal therapy. Previous treatments that are also allowed that do not count as systemic therapy include: surgical resection, transarterial embolization/chemoembolization (TAE/TACE), radiofrequency ablation (RFA), percutaneous ethanol injection (PEI), provided that the lesion(s) to be evaluated in this study are separate from the previously treated lesions(s). Any prior therapy must have been completed >/= 30 days prior to study entry.
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 2.
5. Childs-Pugh status of A or B.
6. Organ function: Absolute peripheral granulocyte count of >/= 1500 mm(3), platelet count of >/= 40,000 mm(3), hemoglobin >/= 10 gm/dL. Total bilirubin </= 2.0 gm/dL; serum albumin >/= 2.5 gm/dL; transaminases up to 5 times the upper limit of institutional normal; and prothrombin time prolonged not more than 3 seconds greater than institutional normal, once attempts to correct a prolonged PT have been made. Patients who require full dose anticoagulation, who are otherwise eligible for this trial, are allowed to have an appropriately prolonged International Normalized Ratio (INR).
7. Negative pregnancy test in women with childbearing potential (those who are not surgically sterilized or who are not amenorrheic for >/= 12 months), within one week prior to initiation of treatment.
8. Fertile men and women must agree to use adequate contraception prior to study entry and for the duration of study participation.
9. Age >/= 18 years. The agents Avastin and erlotinib have not been studied in pediatric patients, thus the doses to be used in this study cannot be assumed to be safe in children.

Exclusion Criteria:

1. Patients who have had prior vascular endothelial growth factor (VEGF) - or epidermal growth factor receptor (EGFR)-targeted therapy.
2. History of prior malignancy other than non-melanoma skin cancer or cervical dysplasia, within five years prior to protocol entry.
3. History of ruptured Hepatocellular carcinoma (HCC) lesion, or HCC lesion with large necrotic areas seen on conventional imaging studies, as determined by the Principal Investigator.
4. Abnormalities of the cornea based on history (eg dry eye syndrome, Sjogren's syndrome) or congenital abnormality (eg Fuch's dystrophy).
5. Gastrointestinal disease resulting in an inability to take oral medication or a requirement for intravenous hyperalimentation.
6. Uncontrolled intercurrent illness including but not limited to: ongoing or active infection requiring parenteral therapy; known HIV disease, New York Heart Association Class II or greater heart failure, cardiac arrhythmia not controlled by medication, uncontrolled psychiatric illness, a history of or current evidence of unexplained nephrotic syndrome, history of uncontrolled hypertension (defined as systolic blood pressure >140 and/or diastolic blood pressure > 90) that is refractory to medical management.
7. Patients may not have received any other investigational agents nor have received any systemic chemotherapy </=30 days prior to enrollment.
8. History of significant gastrointestinal bleeding requiring procedural intervention (eg variceal banding, TIPS procedure, arterial embolization) within 3 months prior to study enrollment. Patients at risk for varices (based on the following: known history of esophageal or gastric varices; evidence of hepatic cirrhosis and/or portal hypertension including biopsy-proven cirrhosis, hypersplenism, or radiographic findings of varices) will be screened for esophageal varices. If varices are identified that require intervention (banding),patient will not be eligible until varices adequately treated.
9. History of myocardial infarction or unstable angina within 6 months.
10. History of stroke within 6 months.
11. Any prior history of hypertensive crisis or hypertensive encephalopathy.
12. Significant or symptomatic vascular disease (e.g., aortic aneurysm, aortic dissection, or peripheral vascular disease).
13. Evidence of clinically significant (Common Toxicity Criteria (CTC) Grade 3 or 4) venous or arterial thrombotic disease within previous 6 months.
14. Current evidence of bleeding disorder or coagulopathy that is not controlled by conservative medical management.
15. Known presence or clinical evidence of central nervous system or brain metastases.
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
17. Minor surgical procedures, fine needle aspirations or core biopsies, excluding placement of a vascular access device, within 7 days prior to Day 0.
18. Pregnant (positive pregnancy test) or lactating.
19. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
20. Serious, non-healing wound, ulcer, or bone fracture.
21. Proteinuria at screening as demonstrated by either: Urine protein:creatinine (UPC) ratio >/= 1.0 at screening, or: Urine dipstick for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
22. Known hypersensitivity to any component of Avastin
23. Inability to comply with study and/or follow-up procedures.
24. Radiographic evidence of major tumor thrombus in the vena cava.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kaseb, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 30, 2005 to May 12, 2009. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 62 participants, three (3) were excluded prior to treatment and are excluded from the trial.
Period: Overall Study
Arm/Group | Bevacizumab + Erlotinib
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 59
Age Continuous [Median (Full Range); unit: years] | 63 [29 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate
Description: Progression free survival (PFS) at 16 weeks of treatment with the combination of Avastin and erlotinib where participant said to be failure free at 16 weeks if they are alive, and their disease has not progressed. PFS Rate is number of participants with PFS at 16 weeks out of total participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline to 16 weeks
Population: Six participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 53
percentage of participants | 64 [51 to 76]

ADVERSE EVENTS:
Time Frame: 3 years and 6 months
Arm/Group | Bevacizumab + Erlotinib
Serious Adverse Events (participants affected / at risk) | 18/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Erlotinib (N=59)
Diarrhea (Gastrointestinal disorders) | 10
Elevated transaminases (Blood and lymphatic system disorders) | 7
Fatigue (General disorders) | 18
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 6
Hypertension (Blood and lymphatic system disorders) | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Erlotinib (N=59)
Abdominal pain (General disorders) | 20
Acne-rash (Skin and subcutaneous tissue disorders) | 22
Anorexia (Gastrointestinal disorders) | 28
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 19
Elevated ALT, AST and bilirubin (Hepatobiliary disorders) | 7 — Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
Fatigue (General disorders) | 18
Hemorrhage, Gastrointestinal (Gastrointestinal disorders) | 3
Low hemoglobin (Blood and lymphatic system disorders) | 3
Mucositis (Gastrointestinal disorders) | 20
Nail changes (Skin and subcutaneous tissue disorders) | 14
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
allergic rhinitis (Immune system disorders) | 7
alopecia (Skin and subcutaneous tissue disorders) | 13
back pain (Musculoskeletal and connective tissue disorders) | 9
dermatology/other (Skin and subcutaneous tissue disorders) | 8
dry eye (Eye disorders) | 25
dry mouth (Gastrointestinal disorders) | 33
dry skin (Skin and subcutaneous tissue disorders) | 37
headache (General disorders) | 20
heartburn (Gastrointestinal disorders) | 11
hemorrhage, pulmonary (Respiratory, thoracic and mediastinal disorders) | 39
hemorrhage, rectum (Gastrointestinal disorders) | 11
hypomagnesemia (Metabolism and nutrition disorders) | 21
insomnia (Psychiatric disorders) | 15
joint pain (Musculoskeletal and connective tissue disorders) | 8
muscle pain (Musculoskeletal and connective tissue disorders) | 15
pruritis (Skin and subcutaneous tissue disorders) | 9
rash-desquamation (Skin and subcutaneous tissue disorders) | 8
rigors/chills (General disorders) | 9
taste alteration (Gastrointestinal disorders) | 18
voice changes (Respiratory, thoracic and mediastinal disorders) | 9
weight loss (Gastrointestinal disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No